CLINICAL TRIAL: NCT06000748
Title: NEPH-ROSIS (NEPHrology in CirRhOSIS) Pilot Trial: A Trial to Treat Acute Kidney Injury Among Hospitalized Cirrhosis Patients
Acronym: NEPH-ROSIS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Investigator Left Institution
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-39806
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Cirrhosis; Portal Hypertension; Hepatorenal Syndrome; Acute Tubule Necrosis; Prerenal Failure
Keywords: PRAGMATIC; FEASIBILITY
MeSH Terms: conditions — Acute Kidney Injury; Fibrosis; Hypertension, Portal; Hepatorenal Syndrome; Kidney Cortex Necrosis

STUDY DESIGN:
Intervention Model Description: This is a single-blind, randomized control, parallel-group, pragmatic trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is single blind. The participants will be blinded to their intervention arm. The treating providers will not be blinded as they will receive either the low or high MAP-target treatment algorithm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low MAP-Target (Active Comparator): This group will be randomized to a treatment algorithm that utilizes a low MAP-target (<80 mmHg) to determine if titration of vasoconstrictors is needed.
  Interventions: Drug: MAP-Target Algorithm
- High MAP-Target (Active Comparator): This group will be randomized to a treatment algorithm that utilizes a high MAP-target (≥80 mmHg) to determine if titration of vasoconstrictors is needed.
  Interventions: Drug: MAP-Target Algorithm

INTERVENTIONS:
Drug: MAP-Target Algorithm — This is a clinical treatment algorithm that will determine the escalation and deescalation of vasoconstrictor utilization based on a target MAP, either high (≥80 mmHg) in the treatment group and low (< 80 mmHg) in the comparator group.

SUMMARY:
The goal of this pilot, randomized, single-blind clinical trial is to estimate the effect size of a high and low mean arterial pressure (MAP)-target algorithm among cirrhosis patients hospitalized with acute kidney injury. The main aims to answer are: • Does an algorithm that has low (<80 mmHg) and high (≥80) MAP-targets lead to significant differences in mean arterial pressure? • Are there any serious adverse events (e.g., ischemia) in a high blood pressure algorithm as compared to a low blood pressure algorithm? • Are there any differences in the incidence of AKI reversal in the high v. low MAP-target groups? Participants will be: 1) Randomized to a clinical algorithm that will either target a low (<80 mmHg) or high (≥80 mmHg) MAP. 2) Depending on their group, investigators will titrate commonly used medications to a specific MAP target. Researchers will compare the high and low MAP-target groups to see if these algorithms lead to significant changes in MAP, if they have any impact on AKI reversal, and if there are any adverse events in the high MAP-target group.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with decompensated cirrhosis, defined as a Child-Pugh Score ≥ 7
* Acute Kidney Injury: a ≥50% increase in sCr from an outpatient baseline sCr measured 7 to 365 days prior to admission

Exclusion Criteria:

1. Patients without a baseline (7 - 365 days prior to AKI development) sCr measurement;
2. Patients who are already on kidney replacement therapy (KRT) at the time of enrollment;
3. Patients with an oxygen requirement greater than 6L via nasal cannula;
4. Patients with a serum creatinine level exceeding 5 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 6 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Differences in mean arterial pressure. | 14 days.
  The investigators will determine if a high, as compared to a low, MAP-target algorithm leads to significantly different changes in MAP. This will be completed by comparing the change in MAP from the baseline to the completion of the study.

SECONDARY OUTCOMES:
Acute kidney injury reversal. | 14 days
  The investigators will determine if a high, as compared to a low, MAP-target algorithm leads to significantly different incidences of acute kidney injury reversal. This will be defined as a decrease in serum creatinine (sCr) to within 0.3 mg/dL of the baseline sCr.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cullaro, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No